CLINICAL TRIAL: NCT01413425
Title: Smith-Lemli-Opitz Syndrome: A Longitudinal Clinical Study of Patients Receiving Cholesterol Supplementation
Brief Title: A Long-Term Study of Cholesterol Supplements for Smith-Lemli-Opitz Syndrome
Status: Withdrawn | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110194; 11-CH-0194
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2014-10-20

CONDITIONS: Smith-Lemi-Opitz Syndrome
Keywords: Smith-Lemli-Opitz Syndrome; Cholesterol; SLOS
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Smith-Lemli-Opitz syndrome (SLOS) is a genetic disorder that prevents the body from making enough cholesterol. People who have SLOS often need to take extra cholesterol, either in food or in supplements, for their bodies to work properly. Cholesterol is very important for the brain and nervous system. Therefore SLOS is highly related to autism, mental retardation, and other brain and nervous system disorders. Not much is known about how people with SLOS handle cholesterol and how taking extra cholesterol helps them. A long-term study of people with SLOS will help answer these and other questions.

Objectives:

- To study the effects of a high-cholesterol diet on people with Smith-Lemli-Opitz syndrome.

Eligibility:

- Individuals of any age who have Smith-Lemli-Opitz syndrome.

Design:

* Participants will have study visits up to two times in the first year and once a year every year after that. Each visit will last between 3 and 5 days.
* Participants will be screened with a physical exam, medical history, and blood and urine tests.
* Participants will provide regular blood, urine, stool, saliva, and skin cell samples for testing.
* Participants will keep track of the foods they eat at home. During the study, they will eat a high-cholesterol diet at all times, except for the second study visit (3 to 6 months after the screening visit). That visit will involve a cholesterol-free diet for 4 weeks.
* Participants will have special cholesterol tests with blood samples at different times during the study.
* At different study visits, participants will have tests of mental and physical skills (including tests for autism). They will answer questions about their diet and food habits. They will also have hearing and eye tests, body and bone measurements, and imaging studies. Not all of the tests will be done at every study.
* Participants will be allowed to leave the study at any time.

DETAILED DESCRIPTION:
The purpose of this study is to learn as much as possible about Smith-Lemli-Opitz Syndrome (SLOS) by following a large group of individuals with SLOS over a period of time. We plan to measure cholesterol and other sterol levels, perform clinical observations, whole body testing and imaging studies (brain MRIs), to learn more about disease mechanisms and progression, variations in the clinical features among individuals with SLOS, and evaluate the effect of cholesterol supplementation in this condition.

Smith-Lemli-Opitz syndrome (SLOS) is a disorder of cholesterol synthesis, or production. It is caused by mutations in the DHCR7 gene which encodes for 7-dehydrocholesterol reductase, an enzyme necessary for the production of cholesterol in the body. Affected individuals exhibit multiple malformations and mental retardation. The features of SLOS are thought to be primarily related to cholesterol deficiency and accumulation of cholesterol precursors. However, the clinical phenotype is not well characterized, the biochemical pathogenesis is incompletely understood, and there is no proven therapy for this devastating condition. Thus our primary objective is to better define the clinical and biochemical phenotypes of the disease using a natural history study design. The study will contribute to creating a comprehensive SLOS patient registry, identify biomarkers that can be used for diagnostic testing, screening and outcome measures in future therapeutic trials. All patients with SLOS receive dietary cholesterol supplementation with the hope that cholesterol supplementation will improve the clinical manifestation of the disease. However, there is no evidence supporting a clinical benefit of cholesterol supplementation. Thus a secondary objective of the study is to determine if cholesterol intake correlates with changes in whole body cholesterol homeostasis and clinical end-points.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion of children:

The population being studied is subjects with SLOS. Children will not be excluded, in fact, the majority of subjects being studied will be infants and children. Relatively few adults with SLOS are known. We will continue to recruit subjects of all ages from newborn to adult of both genders.

Inclusion of women:

Women and girls will certainly be included in the study. Women should be equally represented in this study. SLOS is an autosomal recessively inherited condition that affects males and females equally. However, since these disorders are uncommon autosomal-recessively inherited inborn errors of metabolism, STAIR investigators will have limited control over the gender mix of the study population.

Inclusion of Minorities:

As mentioned for gender, STAIR investigators will have limited control over the race and ethnicity mix of the study population. In order to increase the enrollment of minority subjects, with permission, we will inform the national disease support group of our studies so that subjects in other regions of the US with ethnically and racially more diverse populations may be recruited. SLOS seems to be most common in Caucasians. In the current SLOS study at OHSU, only one of the 34 SLOS subjects is Hispanic. There is only 1 report of carriers in Blacks (Nowaczyk, 2001) and only 31 cases reported in a Japanese survey. In Oregon at least, we will advertise the study at local community health clinics where large numbers of Hispanics are seen.

EXCLUSION CRITERIA:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06-29; Study Completion 2014-10-20

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] SMITH DW, LEMLI L, OPITZ JM. A NEWLY RECOGNIZED SYNDROME OF MULTIPLE CONGENITAL ANOMALIES. J Pediatr. 1964 Feb;64:210-7. doi: 10.1016/s0022-3476(64)80264-x. No abstract available. PMID 14119520
- [Background] Cunniff C, Kratz LE, Moser A, Natowicz MR, Kelley RI. Clinical and biochemical spectrum of patients with RSH/Smith-Lemli-Opitz syndrome and abnormal cholesterol metabolism. Am J Med Genet. 1997 Jan 31;68(3):263-9. PMID 9024557
- [Background] Ryan AK, Bartlett K, Clayton P, Eaton S, Mills L, Donnai D, Winter RM, Burn J. Smith-Lemli-Opitz syndrome: a variable clinical and biochemical phenotype. J Med Genet. 1998 Jul;35(7):558-65. doi: 10.1136/jmg.35.7.558. PMID 9678700